CLINICAL TRIAL: NCT03832114
Title: An Open-label, Non-randomized Study on Efficacy, Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of LNP023 in Two Patient Populations With C3 Glomerulopathy
Brief Title: Study on Efficacy and Safety of LNP023 in C3 Glomerulopathy Patients Transplanted and Not Transplanted
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023X2202
Record Dates: First submitted 2019-01-28; First posted 2019-02-06 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Intervention Model Description: The study is an open-label, two cohort non-randomized study evaluating the efficacy, safety, and pharmacokinetics of LNP023 in patients with C3G (Cohort A) and patients who have undergone kidney transplant and have C3G recurrence (Cohort B).
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - no kidney transplant (Experimental): C3G patients who have not received a kidney transplant and have reduced C3 blood levels.
  Interventions: Drug: LNP023
- Cohort B - kidney transplant (Experimental): C3G patients who have received a kidney transplant and have C3G recurrence.
  Interventions: Drug: LNP023

INTERVENTIONS:
Drug: LNP023 — Increasing doses of LNP023 up to 200 mg.

SUMMARY:
The study is an open-label, two cohort non-randomized study evaluating the efficacy, safety, and pharmacokinetics of LNP023 in patients with C3G (Cohort A) and patients who have undergone kidney transplant and have C3G recurrence (Cohort B).

ELIGIBILITY:
Inclusion Criteria for Cohort A and B:

* Written informed consent must be obtained before any assessment is performed
* Male and female patients between the ages of 18 to 65 (inclusive) at screening
* C3G patients wit proteinuria
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* At screening and baseline visits, patients must weigh at least 35 kg
* Supine vital signs should be within the following ranges :

oral body temperature between 35.0-37.5 °C systolic blood pressure, 80-170 mm Hg diastolic blood pressure, 50-105 mm Hg pulse rate, 45 - 100 bpm

.

Inclusion Criteria for Cohort A:

* Estimated GFR (using the CKD-EPI formula) or measured GFR ≥30 mL/min per 1.73 m2 for patients on a maximum recommended or maximum tolerated dose of an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)
* UPCR ≥ 100 mg/mmol (equivalent to ≥ 1 g/24h total urinary protein excretion)
* Prior to entry, all patients must have been on supportive care including a maximally tolerated dose of ACEi or ARB for at least 30 days.

Inclusion Criteria for Cohort B:

* No histological/laboratory/clinical signs of allorejection
* If applicable, induction treatment after allotransplantation needs to be completed >30 days before inclusion.
* Transplantation of a kidney allograft >90 days before inclusion
* Patients need to be on a stable dose of immunosuppressive regimen prior to inclusion. Any approved treatments are allowed for this purpose.

Exclusion Criteria for Cohort A and B:

* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of randomization, or within 30 days, whichever is longer; or longer if required by local regulations
* A history of clinically significant ECG abnormalities,
* Known family history or known presence of long QT syndrome or Torsades de Pointes
* Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of the study
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 1 week after stopping of investigational drug.
* History of immunodeficiency diseases, or a positive HIV test result.
* Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV).
* Patients who cannot receive vaccinations against N. meningitidis, S. pneumoniae, or H. influenzae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Novartis Investigative Site, Iowa City, Iowa, United States
- France (2):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Ranica, BG, Italy
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wong E, Nester C, Cavero T, Karras A, Le Quintrec M, Lightstone L, Eisenberger U, Soler MJ, Kavanagh D, Daina E, Praga M, Medjeral-Thomas NR, Gackler A, Garcia-Carro C, Biondani A, Chaperon F, Kulmatycki K, Milojevic J, Webb NJA, Nidamarthy PK, Junge G, Remuzzi G. Efficacy and Safety of Iptacopan in Patients With C3 Glomerulopathy. Kidney Int Rep. 2023 Sep 22;8(12):2754-2764. doi: 10.1016/j.ekir.2023.09.017. eCollection 2023 Dec. PMID 38106570
- See also: Link to plain language trial summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients (16 patients in Cohort A and 11 patients in Cohort B) were enrolled and treated in the treatment period 1. All 27 patients completed the study and there were no patients who discontinued the study.
Pre-assignment Details: A total of 27 patients (16 patients in Cohort A and 11 patients in Cohort B) were enrolled and treated in the treatment period 1. All 27 patients completed the study and there were no patients who discontinued the study.
Groups:
- Cohort A: Run-In Phase: Cohort A: No kidney transplant. C3G patients who have not received a kidney transplant and have reduced C3 blood levels
- Cohort B: Run-In Phase: Cohort B: kidney transplant. C3G patients who have received a kidney transplant and have C3G recurrence
- Cohort A: Dose Escalation/LNP023 Treatment 200 mg b.i.d: Cohort A - no kidney transplant C3G patients who have not received a kidney transplant and have reduced C3 blood levels
- Cohort B - Dose Escalation/LNP023 Treatment 200 mg b.i.d: Cohort B - kidney transplant C3G patients who have received a kidney transplant and have C3G recurrence
Period: Run-in Phase
Arm/Group | Cohort A: Run-In Phase | Cohort B: Run-In Phase | Cohort A: Dose Escalation/LNP023 Treatment 200 mg b.i.d | Cohort B - Dose Escalation/LNP023 Treatment 200 mg b.i.d
Started | 16 | 11 | 0 | 0
Completed | 16 | 11 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Escalation/200mg b.i.d Treatment
Arm/Group | Cohort A: Run-In Phase | Cohort B: Run-In Phase | Cohort A: Dose Escalation/LNP023 Treatment 200 mg b.i.d | Cohort B - Dose Escalation/LNP023 Treatment 200 mg b.i.d
Started | 0 | 0 | 16 | 11
Completed | 0 | 0 | 16 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For all analysis sets, patients were analyzed according to study drug received for Cohort A and B. Safety analysis set included all patients that received any study drug. PK analysis set included all patients with available PK data and no protocol deviations with relevant impact on PK data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Customized [Median (Full Range); unit: Years] — Age in Years
  Years | 22.0 [18 to 59] | 31.0 [18 to 70] | 24.0 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 10 | 8 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 16 | 9 | 25
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 8 | 24
  Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Change From Baseline in Urine Protein to Creatinine Concentration Ratio (UPCR)
Description: Change in proteinuria assessed by ratio to baseline of UPCR derived from 24h urine collection
Time Frame: Week 12
Population: Pharmacodynamics (PD) Analysis Set 1: number of patients included in the analysis with at least one post-baseline value of the outcome variable
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant
Number analyzed (Participants) | 16
ratio | 0.55 [0.46 to 0.65]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Test type: Other — Log Ratio to Baseline; p = 0.0003, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.55, 80% CI 2-sided [0.46 to 0.65]

2. Primary Outcome: Cohort B: Change From Baseline in C3 Deposit
Description: Histopathological changes in kidney biopsies as assessed by change from baseline in C3 Deposit Score (based on immunofluorescence microscopy)
Time Frame: Week 12
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Percentage change
Arm/Group | Cohort B - Kidney Transplant
Number analyzed (Participants) | 7
Percentage change | -2.50 [-3.75 to -0.75]
Statistical Analysis 1: Comparison: Cohort B - Kidney Transplant; Test type: Other; p = 0.0313, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.50, 80% CI 2-sided [-3.75 to -0.75]

3. Secondary Outcome: Change From Baseline in Urine Protein Creatinine Concentration Ratio (UPCR)
Description: Ratio to baseline UPCR derived from 24 hour urine collection
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 7
ratio | 0.55 [0.46 to 0.65] | 0.79 [0.49 to 1.28]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.0003, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.55, 80% CI 2-sided [0.46 to 0.65]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.4766, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.79, 80% CI 2-sided [0.49 to 1.28]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.0002, Mixed Model of Repeated Measures (MMRM); Mean Difference (Final Values) = 0.59, 80% CI 2-sided [0.51 to 0.69]

4. Secondary Outcome: Change From Baseline in Urine Protein (UP) Excretion
Description: Ratio to baseline UP excretion derived from 24 hour urine collection
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 9
ratio | 0.57 [0.47 to 0.68] | 1.00 [0.75 to 1.33]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.0011, Mixed Model Repeated Measures (MMRM; Mean Difference (Final Values) = 0.57, 80% CI 2-sided [0.47 to 0.68]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.9998, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 1.00, 80% CI 2-sided [0.75 to 1.33]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.0016, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.66, 80% CI 2-sided [0.56 to 0.77]

5. Secondary Outcome: Change From Baseline in Urine Albumin Creatinine Concentration Ratio (UACR) Excretion
Description: Ratio to baseline UACR excretion derived from 24 hour urine collection
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 7
ratio | 0.55 [0.47 to 0.64] | 0.61 [0.30 to 1.27]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p < 0.0001, Mixed Model Repeated Measures (MRM); Mean Difference (Final Values) = 0.55, 80% CI 2-sided [0.47 to 0.64]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.3707, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.61, 80% CI 2-sided [0.30 to 1.27]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.0002, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.60, 80% CI 2-sided [0.51 to 0.71]

6. Secondary Outcome: Change From Baseline Change in Urinary Albumin (UA) Excretion
Description: Ratio to baseline UA excretion derived from 24 hour urine collection
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 9
ratio | 0.57 [0.47 to 0.70] | 0.81 [0.67 to 0.98]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.0018, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.57, 80% CI 2-sided [0.47 to 0.70]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.1632, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.81, 80% CI 2-sided [0.67 to 0.98]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.0040, Mixed Model Repeated Measure (MMRM); Mean Difference (Final Values) = 0.67, 80% CI 2-sided [0.57 to 0.79]

7. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: Effect of LNP023 on estimated glomerular filtration rate (eGFR)
Time Frame: Day 84
Population: as for outcome 1
Measure: Mean (80% Confidence Interval); unit: ml/min
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 9
ml/min | 2.59 [0.12 to 5.06] | -0.61 [-3.36 to 2.15]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.1795, Mixed Model of Repeated Measures (MMRM); Mean Difference (Final Values) = 2.59, 80% CI 2-sided [0.12 to 5.06]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.7763, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = -0.61, 0.7763% CI 2-sided [-3.36 to 2.15]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.3754, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 1.32, 80% CI 2-sided [-0.59 to 3.22]

8. Secondary Outcome: Change From Baseline in Serum Creatinine
Description: The effect of LNP023 on renal function - serum creatinine
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Mean (80% Confidence Interval); unit: mmol/L
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 9
mmol/L | -5.04 [-9.36 to -0.72] | 7.17 [-1.79 to 16.13]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.1364, Mixed Model Repeated Measuers (MMRM); Mean Difference (Final Values) = -5.04, 80% CI 2-sided [-9.36 to -0.72]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.3038, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 7.17, 80% CI 2-sided [-1.79 to 16.13]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.8352, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = -0.77, 80% CI 2-sided [-5.56 to 4.01]

9. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: The effect of LNP023 on renal function - creatinine clearance
Time Frame: Week 12: Day 84
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: mL/min
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 8
mL/min | 1.07 [0.99 to 1.17] | 1.20 [0.83 to 1.72]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 84; Test type: Other; p = 0.2752, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 1.07, 80% CI 2-sided [0.99 to 1.17]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 84; Test type: Other; p = 0.476, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 1.20, 80% CI 2-sided [0.83 to 1.72]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 84; Test type: Other; p = 0.1963, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 1.10, 80% CI 2-sided [1.00 to 1.20]

10. Secondary Outcome: Number of Patients With Hematuria
Description: The effect of LNP023 on renal function - hematuria
Time Frame: Week 12: Day 84
Population: Pharmacodynamics (PD) Analysis Set 1: number of patients included in the analysis with at least one post-baseline value of the outcome variable. n: number of patients in the respective baseline category and post-baseline time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 9
Participants
  Week 12: Day 84: <9 rbc/hpf n (%) | 10 | 3
  Week 12: Day 84: >= 9 to =<50 rbc/hpf n (%) | 0 | 0
  Week 12: Day 84: >50 rbc/hpf n (%) | 0 | 0

11. Secondary Outcome: Change From Baseline in Urine Protein to Creatinine Concentration Ratio (UPCR) First Morning Void
Description: Ratio to baseline of UPCR reduction derived from total cumulative urinary excretion first morning void
Time Frame: Week 9: Day 64
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: ratio
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 15 | 7
ratio | 0.56 [0.48 to 0.65] | 0.99 [0.76 to 1.28]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 64; Test type: Other; p < 0.0001, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.56, 80% CI 2-sided [0.48 to 0.65]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 64; Test type: Other; p = 0.9544, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.99, 80% CI 2-sided [0.76 to 1.28]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 64; Test type: Other; p < .0001, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.64, 80% CI 2-sided [0.56 to 0.72]

12. Secondary Outcome: Change From Baseline in Urine Albumin to Creatinine Concentration Ratio (UACR) First Morning Void
Description: UACR reduction derived from total cumulative urinary excretion first morning void
Time Frame: Week 9: Day 64
Population: as for outcome 1
Measure: Geometric Mean (80% Confidence Interval); unit: g/mol
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 15 | 7
g/mol | 0.59 [0.50 to 0.69] | 0.87 [0.60 to 1.26]
Statistical Analysis 1: Comparison: Cohort A - no Kidney Transplant; Day 64; Test type: Other; p < .0001, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.59, 80% CI 2-sided [0.50 to 0.69]
Statistical Analysis 2: Comparison: Cohort B - Kidney Transplant; Day 64; Test type: Other; p = 0.6209, Mixed Model Repeated Measures (MMRM); Median Difference (Final Values) = 0.87, 80% CI 2-sided [0.60 to 1.26]
Statistical Analysis 3: Comparison: Cohort A - no Kidney Transplant vs Cohort B - Kidney Transplant; Overall- Day 64; Test type: Other; p = 0.0002, Mixed Model Repeated Measures (MMRM); Mean Difference (Final Values) = 0.63, 80% CI 2-sided [0.54 to 0.73]

13. Secondary Outcome: Pharmacokinetics of LNP023 Area Under the Plasma-concentration-time Curve AUClast (AUC)
Description: The area under the plasma concentration-time curve calculated from time zero to the last quantifiable concentration point (hr*ng/mL)
Time Frame: Day 7, Day 14, Day 21, Day 28 (pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h post dose) and Day 36, Day 64 and Day 84 (pre-dose)
Population: PK Analysis Set: all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort A - no Kidney Transplant - LNP023 10mg b.i.d.: C3G patients who have not received a kidney transplant and have reduced C3 blood levels. Patients received 10 mg b.i.d.of LNP023 during the first treatment week (Week 1) of the dose escalation phase
- Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d.: C3G patients who have not received a kidney transplant and have reduced C3 blood levels. Patients received 25 mg b.i.d.of LNP023 during the second treatment week (Week 2) of the dose escalation phase
- Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d.: C3G patients who have not received a kidney transplant and have reduced C3 blood levels. Patients received 100 mg b.i.d. of LNP023 during the third treatment week (Week 3) of the dose escalation phase
- Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d.: C3G patients who have not received a kidney transplant and have reduced C3 blood levels. Patients received 200 mg b.i.d. of LNP023 during the fourth treatment week (Week 4) of the dose escalation phase, and continued receiving 200 mg b.i.d. for additional 8 weeks (Patients received 200 mg b.i.d. of LNP023 a total of 9 weeks).
- Cohort B - Kidney Transplant - LNP023 10mg b.i.d.: C3G patients who have received a kidney transplant and have C3G recurrence. Patients received 10 mg b.i.d.of LNP023 during the first treatment week (Week 1) of the dose escalation phase
- Cohort B - Kidney Transplant - LNP023 25 mg b.i.d.: C3G patients who have received a kidney transplant and have C3G recurrence. Patients received 25 mg b.i.d.of LNP023 during the second treatment week (Week 2) of the dose escalation phase
- Cohort B - Kidney Transplant - LNP023 100 mg b.i.d.: C3G patients who have received a kidney transplant and have C3G recurrence. Patients received 100 mg b.i.d.of LNP023 during the third treatment week (Week 3) of the dose escalation phase
- Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.: C3G patients who have received a kidney transplant and have C3G recurrence. Patients received 200 mg b.i.d.of LNP023 during the fourth treatment week (Week 4) of the dose escalation phase and continued receiving 200 mg b.i.d. for additional 8 weeks (Patients received 200 mg b.i.d. of LNP023 a total of 9 weeks).
Arm/Group | Cohort A - no Kidney Transplant - LNP023 10mg b.i.d. | Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 10mg b.i.d. | Cohort B - Kidney Transplant - LNP023 25 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 100 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.
Number analyzed (Participants) | 15 | 16 | 16 | 15 | 11 | 11 | 11 | 9
hr*ng/mL | 3690 (693) | 5790 (1630) | 13200 (4410) | 20300 (8180) | 4560 (2060) | 7880 (3830) | 19600 (12100) | 28100 (15900)

14. Secondary Outcome: Pharmacokinetics of LNP023 Area Under the Plasma-concentration-time Curve AUCtau (AUC)
Description: The area under the plasma concentration-time curve calculated to the end of the dosing interval (hr*ng/mL)
Time Frame: Day 7, Day 14, Day 21, Day 28 (pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h post dose) and Day 36, Day 64 and Day 84 (pre-dose)
Population: PK Analysis Set: all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort A - no Kidney Transplant - LNP023 10mg b.i.d. | Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 10mg b.i.d. | Cohort B - Kidney Transplant - LNP023 25 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 100 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.
Number analyzed (Participants) | 15 | 16 | 16 | 15 | 11 | 11 | 11 | 9
hr*ng/mL | 5020 (1110) | 7970 (2250) | 17800 (5800) | 26900 (10900) | 6300 (3000) | 10700 (5310) | 26600 (16500) | 37700 (22000)

15. Secondary Outcome: Observed Maximum Concentration After Drug Administration (Cmax)
Description: The observed maximum plasma concentration (ng/mL)
Time Frame: Day 7, Day 14, Day 21, Day 28 (pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h post dose) and Day 36, Day 64 and Day 84 (pre-dose)
Population: PK Analysis Set: all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A - no Kidney Transplant - LNP023 10mg b.i.d. | Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 10mg b.i.d. | Cohort B - Kidney Transplant - LNP023 25 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 100 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.
Number analyzed (Participants) | 15 | 16 | 16 | 15 | 11 | 11 | 11 | 9
ng/mL | 637 (97.1) | 941 (278) | 2270 (805) | 3600 (1230) | 713 (292) | 1280 (552) | 3250 (1790) | 4700 (2200)

16. Secondary Outcome: Observed Minimum Concentration After Drug Administration (Ctrough)
Description: The concentration that is just prior to the beginning of, or at the end, of a dosing interval (ng/mL)
Time Frame: Day 7, Day 14, Day 21, Day 28 (pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h post dose) and Day 36, Day 64 and Day 84 (pre-dose)
Population: PK Analysis Set: all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A - no Kidney Transplant - LNP023 10mg b.i.d. | Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 10mg b.i.d. | Cohort B - Kidney Transplant - LNP023 25 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 100 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.
Number analyzed (Participants) | 15 | 16 | 16 | 15 | 11 | 11 | 11 | 9
ng/mL | 314 (133) | 519 (133) | 1090 (408) | 1480 (653) | 417 (237) | 644 (325) | 1650 (1010) | 2180 (1610)

17. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax)
Description: The time to reach peak or maximum concentration (hr)
Time Frame: Day 7, Day 14, Day 21, Day 28 (pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h post dose) and Day 36, Day 64 and Day 84 (pre-dose)
Population: PK Analysis Set: all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort A - no Kidney Transplant - LNP023 10mg b.i.d. | Cohort A - no Kidney Transplant - LNP023 25 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 100 mg b.i.d. | Cohort A -no Kidney Transplant - LNP023 200 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 10mg b.i.d. | Cohort B - Kidney Transplant - LNP023 25 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 100 mg b.i.d. | Cohort B - Kidney Transplant - LNP023 200 mg b.i.d.
Number analyzed (Participants) | 15 | 16 | 16 | 15 | 11 | 11 | 11 | 9
hr | 2.00 [0.800 to 6.00] | 2.00 [0.900 to 4.00] | 2.00 [0.500 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00]

18. Secondary Outcome: Summary of Change From Baseline Complement C3 Biomarker in Serum
Description: To assess the effect of LNP023 on alternative complement pathway hyperactivity.
Time Frame: Baseline, Day 1, Day 7, Day 14, Day 21, Day 28, Day 36, Day 64, Day 84
Population: PD Analysis Set 2: included all patients with available Pharmacodynamics (PD) data and no protocol deviations with relevant impact on PD data. At each timepoint only subjects with a value at both baseline and that timepoint were included.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 10
g/L
  Day 1 pre-dose | 0.0 (0.06) | 0.0 (0.12)
  Day 7 - pre-dose | 0.1 (0.10) | 0.2 (0.22)
  Day 14 - pre-dose | 0.3 (0.17) | 0.4 (0.29)
  Day 21 - pre-dose | 0.5 (0.25) | 0.4 (0.33)
  Day 28 - pre-dose: number analyzed (Participants) | 15 | 9
  Day 28 - pre-dose | 0.5 (0.29) | 0.4 (0.27)
  Day 36 - pre-dose: number analyzed (Participants) | 16 | 9
  Day 36 - pre-dose | 0.6 (0.28) | 0.4 (0.32)
  Day 64 - pre-dose: number analyzed (Participants) | 15 | 8
  Day 64 - pre-dose | 0.6 (0.27) | 0.4 (0.26)
  Day 84 - pre-dose | 0.6 (0.30) | 0.5 (0.26)

19. Secondary Outcome: Ratio to Baseline Summary of Plasma Bb
Description: To assess the relationship between LNP023 dose and pharmacodynamic biomarker levels of blood Bb
Time Frame: Baseline, Day 1, Day 7, Day 14, Day 21, Day 28, Day 36, Day 64, Day 84
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Ratio of plasma Bb
Arm/Group | Cohort A - no Kidney Transplant | Cohort B - Kidney Transplant
Number analyzed (Participants) | 16 | 10
Ratio of plasma Bb
  Day 1 pre-dose: number analyzed (Participants) | 15 | 10
  Day 1 pre-dose | 101.8 (45.18) | 109.7 (34.08)
  Day 7 pre-dose: number analyzed (Participants) | 15 | 10
  Day 7 pre-dose | 102.4 (40.47) | 83.6 (27.73)
  Day 14 pre-dose | 104.4 (43.35) | 81.8 (39.34)
  Day 21 pre-dose | 97.0 (58.06) | 66.4 (22.95)
  Day 28 pre-dose: number analyzed (Participants) | 15 | 9
  Day 28 pre-dose | 90.2 (46.24) | 71.5 (29.52)
  Day 36 pre-dose: number analyzed (Participants) | 16 | 9
  Day 36 pre-dose | 102.5 (54.06) | 65.9 (31.20)
  Day 64 pre-dose: number analyzed (Participants) | 15 | 8
  Day 64 pre-dose | 116.8 (59.76) | 73.2 (29.62)
  Day 84 pre-dose | 116.6 (57.85) | 76.3 (35.84)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 2 years, 2 months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- Cohort A - Run-in Phase; Cohort A - Dose Escalation Phase; Cohort A - LNP023 200mg b.i.d: No Kidney Transplant- C3G patients who have not received a kidney transplant and have reduced C3 blood levels
- Cohort B - Run-in Phase; Cohort B - Dose Escalation Phase; Cohort B - LNP023 200mg b.i.d: Kidney Transplant- C3G patients who have received a kidney transplant and have C3G recurrence
Arm/Group | Cohort A - Run-in Phase | Cohort A - Dose Escalation Phase | Cohort A - LNP023 200mg b.i.d | Cohort B - Run-in Phase | Cohort B - Dose Escalation Phase | Cohort B - LNP023 200mg b.i.d
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/11 | 0/11 | 2/11
Other Adverse Events (participants affected / at risk) | 0/16 | 6/16 | 8/16 | 0/11 | 5/11 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Run-in Phase (N=16) | Cohort A - Dose Escalation Phase (N=16) | Cohort A - LNP023 200mg b.i.d (N=16) | Cohort B - Run-in Phase (N=11) | Cohort B - Dose Escalation Phase (N=11) | Cohort B - LNP023 200mg b.i.d (N=11)
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Run-in Phase (N=16) | Cohort A - Dose Escalation Phase (N=16) | Cohort A - LNP023 200mg b.i.d (N=16) | Cohort B - Run-in Phase (N=11) | Cohort B - Dose Escalation Phase (N=11) | Cohort B - LNP023 200mg b.i.d (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Blood luteinising hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Spider vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT03832114/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03832114/SAP_001.pdf